CLINICAL TRIAL: NCT06875674
Title: Selenium Biofortification of Strawberries and Human Intervention
Brief Title: Selenium Biofortification of Strawberries
Acronym: SeStra30Days
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Sara Baldassano, Professor, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SeStraw30Days24
Record Dates: First submitted 2025-03-07; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Nutrition, Healthy
MeSH Terms: interventions — Dietary Supplements; Selenium; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Placebo Comparator): The control group received strawberries (control strawberries 100grams/day) that was without biofortification with the same characteristic of strawberries lettuce(soil, water, harvesting time) for 30 days
  Interventions: Dietary Supplement: supplementation with control strawberry
- Selenium-biofortified strawberry supplementation (Active Comparator): This group will received selenium biofortified strawberries (100grams/day) with the same characteristic of control strawberries lettuce(soil, water, harvesting time) for 30 days
  Interventions: Dietary Supplement: supplementation with biofortified strawberry
- Tablet Selenium supplementation (Active Comparator): This group will received selenium in tablet (100 micrograms/day) for 30 days
  Interventions: Dietary Supplement: supplementation with selenium in tablet

INTERVENTIONS:
Dietary Supplement: supplementation with control strawberry — control strawberry supplementation (100 grams/day) for 30 days
  Arms: Control group
Dietary Supplement: supplementation with biofortified strawberry — selenium biofortified strawberry supplementation (100 grams/day) for 30 days
  Arms: Selenium-biofortified strawberry supplementation
Dietary Supplement: supplementation with selenium in tablet — selenium supplementation in tablet (100 micrograms/day) for 30 days
  Arms: Tablet Selenium supplementation

SUMMARY:
This study aims to investigate the effects of a nutritional intervention with selenium-biofortified strawberries on glucose homeostasis and hepatic function of healthy individuals. The study will assess if consumption of selenium-biofortified strawberries would increase the selenium endogenous concentration (primary outcome) and if it would impact, and to which extension, glucose homeostasis and hepatic function (secondary outcome).

DETAILED DESCRIPTION:
Selenium is an essential micronutrient with antioxidant properties and a crucial role in various physiological processes. Biofortification of crops with selenium offers a promising strategy to enhance selenium intake and improve human health. Strawberries are a widely consumed fruit and can serve as an effective vehicle for selenium delivery. The effects of consuming selenium-biofortified strawberries on human health will be investigated.

3. Study Goals and Objectives

The primary objective is to evaluate the impact of consuming selenium-biofortified strawberries for 30 days on serum selenium concentration in healthy adults. The secondary objective is to assess the influence of this intervention on glucose profile and hepatic function. • Fifty-five healthy adult volunteers (both sexes) will be randomly assigned to three groups:

* Control group: Consuming 100 grams of control strawberries daily.
* Intervention group (selenium-biofortified strawberries): Consuming 100 grams of selenium-biofortified strawberries daily.
* Intervention group (selenium supplement): Consuming a selenium supplement of 100 micrograms daily.

  * The intervention period will be 30 days.
  * Blood samples (serum and plasma) will be collected at baseline (T0) and at the end of the intervention (T30).
  * Body weight, barefoot standing height, body mass index, and body composition will be measured at baseline and T30.
  * Blood samples will be analyzed for:
* Selenium.
* Glucose
* Insulin
* insulin resistance
* insulin sensitivity
* β-cell function
* aminotransferase (AST)
* alanine aminotransferase (ALT)
* gamma-glutamyl transferase (GGT)
* albumin (ALB)

  * Data will be recorded in a coded database to ensure participant privacy.
  * Samples will be transported in certified containers for biological samples, and processed at the Molecular Biology section of the University of Palermo.

The statistical analyses will be carried out using specific software. To compare the baseline characteristics of the groups student t tests will be used. The comparison between the different groups of participants and within the same group between baseline and T30 will be carried out using One-Way ANOVA followed by Sidak test. Values will be expressed as mean ± standard deviation (mean ± SD). P-value ≤ 0.05 will be considered to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 - 65 years
* Italian Ethnicity
* Body mass index between 18.5 and 28.5 kg/m²
* Clinically Healthy

Exclusion Criteria:

* Chronic disease
* Use of drugs (excluding occasional over the counter medications)
* Pregnancy
* Exogenous hormone use
* Breastfeeding
* Use of supplements

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-03-07 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-09-29 (Actual)

PRIMARY OUTCOMES:
Measurement of selenium concentration in participants | 30 days
  Selenium (μg/L) will be measured in serum at baseline and after 30 days

SECONDARY OUTCOMES:
Measurement of glucose in participants | 30 days
  Glucose (mg/dL) will be measured in serum at baseline and after 30 days
Measurement of insulin in participants | 30 days
  Insulin (mUI/L) will be measured in serum at baseline and after 30 days
Measurement of insulin resistance in participants | 30 days
  Insulin resistance (HOMA-IR) will be calculated from fasting glucose and insulin levels at baseline and after 30 days
Measurement of insulin sensitivity in participants | 30 days
  Insulin sensitivity (QUICKI) will be calculated from fasting glucose and insulin levels at baseline and after 30 days
Measurement of β-cell function in participants | 30 days
  β-cell function (HOMA-β) will be calculated from fasting glucose and insulin levels at baseline and after 30 days
Measurement of aminotransferase (AST) in participants | 30 days
  AST (U/L) will be measured in serum at baseline and after 30 daysbaseline and after 30 days
Measurement of alanine aminotransferase (ALT) in participants | 30 days
  ALT (U/L) will be measured in serum at baseline and after 30 days
Measurement of gamma-glutamyl transferase (GGT) in participants | 30 days
  GGT (U/L) will be measured in serum at baseline and after 30 days
Measurement of albumin (ALB) in participants | 30 days
  ALB (g/dL) will be measured in serum at baseline and after 30 days

OTHER OUTCOMES:
Measurement of Height in participants | baseline
  Height (meters) will be assessed at baseline
Measurement of body weight in participants | 30 days
  Body weight (kg) will be assessed at baseline and after 30 days
Measurement of body mass index (BMI) in participants | 30 days
  Weight in kilograms, height in meters will be aggregated to arrive at one reported value (weight and height will be combined to report BMI in kg/m²)
Measurement of body composition in participants | 30 days
  Lean mass as percent of body weight and fat mass as percent of body weight will be assessed at baseline and after 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Sara Baldassano, Principal Investigator — NABbio, STEBICEF department Palermo, Italy, 90128
Locations (1):
- Department of Biological, Chemical and Pharmaceutical Sciences and Technologies, Palermo University, Palermo, PA, Italy